CLINICAL TRIAL: NCT03158935
Title: Phase Ib Trial of Pembrolizumab Administered in Combination With or Following Adoptive Cell Therapy- A Multiple Cohort Study; The ACTIVATE (Adoptive Cell Therapy InVigorated to Augment Tumor Eradication) Trial
Brief Title: The ACTIVATE (Adoptive Cell Therapy InVigorated to Augment Tumor Eradication) Trial
Acronym: ACTIVATE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTIVATE
Record Dates: First submitted 2017-05-09; First posted 2017-05-18 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Advanced Ovarian Cancer; Malignant Melanoma
Keywords: adoptive cell therapy; melanoma; ovarian; cyclophosphamide; fludarabine; tumor-infiltrating lymphocytes (TILs); pembrolizumab; interleukin-2; anti-PD-1; immune checkpoint
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; pembrolizumab; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Advanced metastatic melanoma (Cohort 1) (Experimental): Cyclophosphamide and fludarabine followed by Tumor-Infiltrating Lymphocytes (TILs), Interleukin-2 (IL-2), and pembrolizumab
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Pembrolizumab; Biological: Tumor-Infiltrating Lymphocytes (TILs); Biological: Interleukin-2 (IL-2)
- Advanced ovarian cancer (Cohort 2): (Experimental): Cyclophosphamide followed by Tumor-Infiltrating Lymphocytes (TILs), Interleukin-2 (IL-2), and pembrolizumab
  Interventions: Drug: Cyclophosphamide; Procedure: Pembrolizumab; Biological: Tumor-Infiltrating Lymphocytes (TILs); Biological: Interleukin-2 (IL-2)

INTERVENTIONS:
Drug: Cyclophosphamide — Cohort 1: i.v., 60mg/kg per day for 2 days Cohort 2: i.v., 30mg/kg per day for 2 days
  Other Names: Cytoxan, Procytox
Drug: Fludarabine — Cohort 1: i.v., 25mg/m2 per day for 5 days
  Other Names: Fludara
  Arms: Advanced metastatic melanoma (Cohort 1)
Procedure: Pembrolizumab — Cohort 1 and 2: i.v., 200mg every 3 weeks
  Other Names: Keytruda, MK-3475
Biological: Tumor-Infiltrating Lymphocytes (TILs) — Cohort 1 and 2: i.v., 1x10^10 - 1.6x10^11 cells
Biological: Interleukin-2 (IL-2) — Cohort 1 and 2: i.v., 125,000 IU/kg subcutaneous per day
  Other Names: Aldesleukin, Proleukin, Recombinant Human Interleukin 2

SUMMARY:
This is a phase 1b study for patients with metastatic (cancer has spread to various parts of the body) melanoma and ovarian cancer. The main purpose is to examine the safety and efficacy of administering pembrolizumab after receiving chemotherapy, tumor-infiltrating lymphocytes (TIL) and low dose interleukin 2 (IL-2).

Patients will first receive either cyclophosphamide, or cyclophosphamide and fludarabine. These are chemotherapy agents that prepare the body to receive TILs.

Patients are then infused with autologous TILs, a type of white blood cell that recognizes tumor cells and enters them, thereby causing tumor cells to break down.

Following TILs infusion, patients will receive low-dose IL-2 therapy. This is a type of protein that is intended to activate and stimulate the growth of cells in the patient's immune system.

If the patient meets the required criteria, they will be given pembrolizumab, a monoclonal antibody (drug made up of cloned immune cells) that is designed to block a protein called programed cell death ligand 1 (PD-L1) which will allow the body's immune system to kill the cancer cells.

DETAILED DESCRIPTION:
This study will involve treatment with chemotherapy, TILs, IL-2, pembrolizumab, tests and procedures done for safety, and the collection of archival tumor tissue, fresh tumor biopsies, and blood samples for biomarker research.

ELIGIBILITY:
Pre-TIL Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Have measurable disease based on RECIST 1.1.
4. Have a performance status of 0 or 1 on the ECOG Performance Scale.
5. Demonstrate adequate organ function, all screening labs should be performed within 10 days of treatment initiation.
6. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
7. Female subjects of childbearing potential must be willing to use an adequate method of contraception - Contraception, for the course of the study through 6 months after the last dose of cyclophosphamide or fludarabine, or 120 days after last dose of pembrolizumab, whichever is longer.
8. Male subjects of childbearing potential must agree to use an adequate method of contraception - Contraception, starting with the first dose of study therapy through 6 months after the last dose of cyclophosphamide or fludarabine, or 120 days after last dose of pembrolizumab, whichever is longer.

Cohort 1 Pre-TIL inclusion criteria:

1. Metastatic melanoma with surgically unresectable stage III or stage IV, histologically confirmed
2. Previously treated with anti-PD-1 or anti-PD-L1 therapy (such as pembrolizumab or nivolumab) and experienced progression by RECIST v1.1
3. Prior systemic anti-CTLA-4 therapy is allowed, provided that the first dose of pembrolizumab on study is administered more than 6 weeks after the last dose of anti-CTLA-4 treatment.
4. Progression of disease by RECIST 1.1 within 3 months of last dose of therapy. If no alternative standard therapy is available, and there is evidence of clinical progression, subjects may proceed with TIL therapy after discussion with the Sponsor.

Cohort 2 Pre-TIL inclusion criteria:

1. Platinum resistant ovarian cancer, histologically confirmed

   • Platinum resistant as defined by evidence of radiographic progression within 6 months of the last dose of platinum.
2. Prior systemic anti-CTLA-4 therapy is allowed, provided that the first dose of pembrolizumab is administered more than 6 weeks after the last dose of anti-CTLA-4 treatment.
3. Eligible for ACT with autologous TIL

Both Cohorts 1 and 2 (pre-TIL):

1. Subjects may have 3 or fewer asymptomatic brain metastases, ≤ 1 cm in size each. Note: If lesions are symptomatic, >1 cm each in size, or more than 3 in number, these lesions must undergo definitive treatment with surgery and/or radiation at least four weeks days prior to the first dose of lymphodepleting chemotherapy. If in the opinion of the PI or his designee the lesion(s) no longer represents active disease, the subject will be considered eligible.
2. No history of serious cardiac illness including (but not confined to):

   * Previous or active myocardial infarction in the past 2 years
   * Congestive cardiac failure (NYHA III or IV)
   * Unstable angina pectoris
   * Recent coronary artery bypass grafting <6 months
   * Uncontrolled hypertension (systolic greater than or equal to 160 mmHg or diastolic greater than or equal to 100 mmHg)
   * Ventricular arrhythmia < 6 months
3. Subjects who have a prolonged history of cigarette smoking or symptoms of respiratory dysfunction should not have abnormal pulmonary function test as evidenced by a FEV1 < 60% predicted within 4 weeks of chemotherapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active, untreated TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy within 28 days prior to study Day 1, or targeted small molecule therapy or radiation therapy within 14 days prior to study Day 1. Patients who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, and in situ cervical cancer that has undergone potentially curative therapy.
8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Has known history of, or any evidence of active, non-infectious pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 6 months after last dose of cyclophosphamide or fludarabine or 120 days after the last dose of pembrolizumab.
14. Has a known history of Human Immunodeficiency Virus (HIV) (e.g. HIV 1/2 antibody positive) or Human T-Cell Lymphotropic Virus (HTLV).
15. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
16. Untreated syphilis.
17. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Subjects with ongoing prior use of systemic steroid therapy within 4 weeks before the TILs infusion will be excluded. Use of topical, intranasal and inhaled corticosteroids, or systemic corticosteroids at physiologic doses are allowed.

Cohort 1 and 2 Post-TIL (pembrolizumab) inclusion criteria:

1. Previously met applicable inclusion and exclusion criteria.
2. Initiation of pembrolizumab therapy must occur more than 21 days after the last dose of fludarabine.
3. Resolution of TIL protocol related adverse events to grade 2 or less. Otherwise, patients may proceed with pembrolizumab therapy if the treating investigator, after discussion with the Sponsor, determines that residual TIL therapy related adverse events are not clinically significant.

Cohort 1 and 2 Post-TIL (pembrolizumab) exclusion criteria:

1. Has an active infection requiring systemic therapy. (Prophylactic antibiotics and antiviral agents are allowed.)
2. Has developed a condition or requires a therapy that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
3. Development of a condition that, in the opinion of the investigator, would be a contraindication for initiating pembrolizumab therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Monitoring of serious adverse events to determine the safety of initiating pembrolizumab following lymphodepleting chemotherapy, TIL administration, and low dose IL-2 injections within 35 days of TIL infusion. | 2 years
  Toxicities will be monitored on an ongoing basis. Severe adverse events will be reviewed for attribution to the study drug and whether they resolve to an acceptable grade within 35 days of TIL infusion. This information will be used to determine if the patient will go on to receive pembrolizumab. The regimen will be deemed feasible if at least 80% of patients enrolled go on to receive pembrolizumab.

SECONDARY OUTCOMES:
Overall Response Rate | 2 years
  To evaluate the response rate of pembrolizumab following or in combination with ACT using measurable disease by RECIST v1.1.
Overall and Progression Free Survival | 2 years
  To evaluate the survival outcomes of overall and progression free survival per tumour type
Safety profile of pembrolizumab therapy given after or in combination with ACT in patients with advanced melanoma and ovarian cancer using CTCAE v4.0 | 2 years
  Events that are both unrelated and related to treatment will be captured using CTCAE v4.0. The total number of episodes for each event will be reported, as well as the severity and attribution to study therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Butler, M.D., Principal Investigator — Tumor Immunotherapy Program, Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No